CLINICAL TRIAL: NCT03300791
Title: Predictive Models of Readmission in Heart Failure: Profile of Readmitted Patients
Brief Title: Predictive Models of Readmission in Heart Failure
Acronym: REIC
Status: Completed | Type: Observational
Sponsor: Hospital Galdakao-Usansolo (Other Government)
Collaborators: Hospital de Basurto (Other); Hospital Donostia (Other); Hospital de Mendaro (Unknown); Hospital Costa del Sol (Other); Corporacion Parc Tauli (Other)
Responsible Party: Principal Investigator, Susana García Gutiérrez, PhD, Hospital Galdakao-Usansolo
Other Study IDs: PI15/01343-2015111003
Record Dates: First submitted 2017-09-26; First posted 2017-10-03 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Heart Failure
Keywords: heart failure; readmission; predictive models
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Admitted: We will include patients who had beeb admitted by an acute heart failure in hospitalization ward
  Interventions: Other: Admitted

INTERVENTIONS:
Other: Admitted — Readmitted patients in the next months after an episode of aute heart failure will be recruited. Controls will be selected between those who were admitted in the baseline but not readmitted in this month.
  Other Names: Not readmitted

SUMMARY:
This is a prospective nested case-control study.

Our goals are to create predictive models to readmissions for heart failure and also to define profiles for patients who are readmitted during the first month after the index episode.

Patients who will be admitted in five hospitals in spain by the reason of a heart failure will be recruited during 18 months. Those who will be readmitted in a hospital up to a month after the index episode will be considered cases. Controls will be selected from the initial cohort of hospitalized patients.

DETAILED DESCRIPTION:
Objective: To create models for predicting the risk of readmission short term (30-90 days) and medium term (one year).To identify differences between patients readmitted and not readmitted, and profiles of frequently preventable readmissions in our setting.

Methodology: Observational prospective cohort of patients who are discharged with a diagnosis of heart failure in 5 participating centers. further, a nested case-control will be developed in the previous cohort, being cases those readmitted and controls will be chosen according to age, sex, etiology of heart failure, comorbidities and functional status. Sociodemographic, clinical and health related quality of life, empowerment and baseline self-efficacy as predictors of readmission were collected.

Regarding the cases and controls, the quality of life in post-discharge transitional period, empowerment and self-efficacy, caregiver burden, social support, discharge care model, use of health services and adequation, conciliation and adherence to treatment will be assessed . Cox proportional hazards models will be created, and conditional logistic regression models to identify differences between cases and controls.

Expected Results: National Health System will be provided with tools for predicting the risk of readmission useful to clinicians and managers to offer discharge individualized care. The most common characteristics of readmissions and preventable readmissions will be identified, which will be helpful to create specific actions in the future.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted by acute heart failure (de novo and acute decompensated) (International Classification of Diseases, Ninth Revision, Clinical Modification: 428.x; some of the 402.x group), older tan 18 who will accept to participate.

Exclusion Criteria:

* patients who develop HF episodes during admission, if have been admitted for another reason,
* patients transferred from other health centers,
* myocardial infarction or stroke in the 4 weeks prior to admission,
* life expectancy less than one year, for HF at the terminal or cause different from the CI according to the assessment of the study subjects,
* inability to complete the questionnaires or with assistance external (reviewer, family, social) because of sensorineural reason, dementia or ignorance of the language.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted by the reason of heart failure
Sampling Method: Non-Probability Sample
Enrollment: 1250 (Actual)
Dates: Start 2017-09-28 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Readmission | 1 month
  Up to a month after admission by heart failure

SECONDARY OUTCOMES:
Readmission | 12 months
  Up to 12 months after admission by heart failure

CONTACTS AND LOCATIONS:
Overall Officials: Susana Garcia-Gutierrez, PhD, Principal Investigator — Unidad de Investigación. Hospital Galdakao-Usansolo. Osakidetza
Locations (4):
- Spain (4):
  - Marisa Bare, Sabadell, Barcelona
  - Ainara, Bilbao, Bizkaia
  - Irene Rilo, Donostia / San Sebastian, Gipuzkoa
  - Raul, Marbella, Málaga

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Garcia-Gutierrez S, Villanueva A, Lafuente I, Rodriguez I, Lozano-Bahamonde A, Murga N, Orus J, Camacho ER, Quintana JM, Quiros R; ReIC-REDISSEC working group. Factors related to early readmissions after acute heart failure: a nested case-control study. BMC Cardiovasc Disord. 2023 Jan 12;23(1):17. doi: 10.1186/s12872-022-03029-2. PMID 36635633